CLINICAL TRIAL: NCT06997016
Title: Enhanced Recovery After Surgery (ERAS) in Live Donor Kidney Transplant Recipients
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Baylor IRB #025-220
Record Dates: First submitted 2025-05-21; First posted 2025-05-30 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-05

CONDITIONS: Postoperative Pain
Keywords: transplantation, kidney; renal transplantation; Enhanced Postsurgical Recovery; Recovery, Enhanced Postsurgical; pain, postoperative; postsurgical pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Gabapentin; Bupivacaine; Walking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Enhanced Recovery Protocol (Experimental): This group will receive the following:
  50g carbohydrate drink 2 hours prior to surgery 300mg of gabapentin 30 minutes prior to surgery 650mg of acetaminophen 30 minutes prior to surgery 0.25% bupivicaine local anesthetic intraoperatively assisted ambulation 12 hours after surgery
  Interventions: Dietary Supplement: pre-operative carbohydrate drink; Drug: Acetaminophen; Drug: Gabapentin; Drug: Bupivacaine; Other: Ambulation
- Control group (No Intervention): This group is a retrospective review of 30 patients who have undergone a live donor kidney transplant during 1/1/2022-12/31/2024 will be selected and undergo a retrospective chart review for the same data collection points.

INTERVENTIONS:
Dietary Supplement: pre-operative carbohydrate drink — 50 g of carbohydrate drink 2 hours before surgery
  Arms: Enhanced Recovery Protocol
Drug: Acetaminophen — 650mg acetaminophen 30 minutes prior to surgery
  Other Names: tylenol
  Arms: Enhanced Recovery Protocol
Drug: Gabapentin — 300 mg gabapentin 30 minutes prior to surgery
  Other Names: Neurontin; Gralise
  Arms: Enhanced Recovery Protocol
Drug: Bupivacaine — intraoperative local anesthetic
  Other Names: Marcaine; Sensorcaine
  Arms: Enhanced Recovery Protocol
Other: Ambulation — Assisted ambulation 12 hours after surgery
  Arms: Enhanced Recovery Protocol

SUMMARY:
The goal of this interventional study is to learn if an Enhanced Recovery After Surgery (ERAS) protocol works to reduce the need for narcotic pain medications in live donor kidney transplant recipients. The main questions it aims to answer are:

Does the ERAS protocol lower the amount of opioid narcotic medication needed to manage post-surgery pain? Does the ERAS protocol help lower pain scores after surgery? Researchers will compare the ERAS protocol to previous patients where the ERAS protocol was not used to see if the ERAS protocol works to reduce post-surgery pain.

Participants will be asked to:

* Drink a pre-surgery carbohydrate drink two hours before your surgery.
* Take a pre-surgery dose of Tylenol by mouth.
* Take a pre-surgery dose of Gabapentin by mouth.
* The surgeon will administer a local numbing medication at the surgery site by injection during the surgery.
* Begin walking with assistance about 12 hours after your surgery.
* Allow the research staff to collect data about your kidney function. This data will be collected on your postoperative clinic visits, which generally occur about twice weekly for one month. This information will determine your kidney health, need for hospitalization, and side effects that may occur.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* over 18 years of age
* receiving a kidney transplant from a living donor.

Exclusion Criteria:

* delayed gastric emptying
* severe type I diabetes
* allergy to interventional medications
* pregnancy (this is a normal exclusion for kidney recipients)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) (0-10) | From enrollment to the end of treatment at 30 days
  Patient reported pain on a scale from 0 (no pain) to 10 (the worst possible pain)
Narcotic Use | From enrollment to the end of treatment at 30 days
  milligram morphine equivalents (MME)

SECONDARY OUTCOMES:
Adverse Events | From enrollment to the end of treatment at 30 days
  unfavorable medical occurence
Hospital readmission | From enrollment to the end of treatment at 30 days
  readmission to any hospital within 30 days
Length of Stay | From enrollment to the end of treatment at 30 days
  total hospital length of stay

CONTACTS AND LOCATIONS:
Overall Officials: Richard Ruiz, MD, Principal Investigator — Baylor Scott & White All Saints Medical Center
Locations (1):
- Baylor Scott & White All Saints Medical Center, Fort Worth, Texas, United States

IPD SHARING:
Plan to Share IPD: No